CLINICAL TRIAL: NCT02398773
Title: [18F] Fluoroestradiol (FES) PET as a Predictive Measure for Endocrine Therapy in Patients With Newly Diagnosed Metastatic Breast Cancer
Brief Title: FES PET/CT in Predicting Response in Patients With Newly Diagnosed Metastatic Breast Cancer Receiving Endocrine Therapy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NCI-2015-00383; NCI-2015-00383 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAI142; PEAI142_R01PAPP01; EAI142 (Other: ECOG-ACRIN Cancer Research Group); EAI142 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2015-03-25; First posted 2015-03-26 (Estimated); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: HER2/Neu Negative; Progesterone Receptor Negative; Progesterone Receptor Positive; Stage IV Breast Cancer AJCC v6 and v7
MeSH Terms: interventions — 16-fluoroestradiol; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (FES PET/CT) (Experimental): Between 0 to 30 days before start of endocrine therapy, patients receive F-18 16 alpha-fluoroestradiol IV over 2 minutes and undergo PET/CT. Patients may undergo a second FES-PET/CT study at least 24 hours after the first study and no later than 10 days after the initial study.
  Interventions: Procedure: Computed Tomography; Drug: F-18 16 Alpha-Fluoroestradiol; Other: Laboratory Biomarker Analysis; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: F-18 16 Alpha-Fluoroestradiol — Given IV
  Other Names: 16 alpha-fluroestradiol-17 beta; F-18 FES; FES; Fluorine-18 16 alpha-fluoroestradiol; Fluoroestradiol F-18
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT

SUMMARY:
This phase II trial studies F-18 16 alpha-fluoroestradiol (FES) positron emission tomography (PET)/computed tomography (CT) in predicting response to endocrine therapy in patients with newly diagnosed breast cancer that has spread to other parts of the body. FES is a radioactive form of the hormone estrogen and may "light up" where cancer is in the body. Diagnostic procedures using FES, such as FES PET/CT, may help measure the FES and help doctors predict how well the cancer will respond to treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the negative predictive value (NPV) of [18F]fluoroestradiol (FES) uptake for response (clinical benefit) at 6 months in patients with estrogen-receptor positive (ER+) metastatic breast cancer treated with first-line endocrine therapy.

SECONDARY OBJECTIVES:

I. To determine the test-retest reproducibility of quantitative assessment of tumor FES uptake by standardized uptake values (SUVs).

II. To evaluate the accuracy of FES-PET/CT for predicting response in patients treated with first line endocrine therapy for metastatic breast cancer.

III. To evaluate the accuracy of FES-PET/CT for predicting progression-free survival (PFS) in patients treated with first line endocrine therapy for metastatic breast cancer.

IV. To examine the role of FES-PET/CT in predicting progressive disease (PD) or clinical benefit (CB), in concert with semi-quantitative interpretation of ER, progesterone receptor (PgR), and marker of proliferation Ki-67 (Ki-67).

V. To evaluate the relationships among FES uptake, as measured by maximum SUV (SUVmax) and semi-quantitative ER from immunohistochemistry (IHC).

VI. To evaluate FES SUVmax < 1.5 as the optimal cutpoint for predicting progression-free survival (PFS) to first line endocrine therapy for metastatic breast cancer.

VII. To determine the percent of eligible patients for whom biopsy is not feasible, i.e., determine the clinical utility of indirect assay of ER expression by FES-PET/CT.

VIII. To evaluate the heterogeneity of tumor FES uptake in individual patients defined as variability in lesion's FES uptake.

OUTLINE:

Between 0 to 30 days before start of endocrine therapy, patients receive F-18 16 alpha-fluoroestradiol intravenously (IV) over 2 minutes and undergo PET/CT. Patients may undergo a second FES-PET/CT study at least 24 hours after the first study and no later than 10 days after the initial study.

After completion of study, patients are followed up for 6 months and then periodically for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Capable and willing to provide informed consent
* Women must not be pregnant or breast-feeding. All females of childbearing potential must have a blood test or urine study within 7 days prior to FES PET/CT scan and [18F]-fluorodeoxyglucose (FDG)-PET/CT scan to rule out pregnancy; a female of childbearing potential is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria:

  * Has not undergone a hysterectomy or bilateral oophorectomy or
  * Has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Women of childbearing potential and sexually active males must use an accepted and effective method of contraception or to abstain from sexual intercourse for the duration of their participation in the study
* Patient is a postmenopausal woman, man, or premenopausal woman for whom standard endocrine therapy alone (tamoxifen, aromatase inhibitor [AI], with or without ovarian suppression or fulvestrant) is planned after FES-PET/CT is completed
* Medically stable as judged by patient's physician
* Life expectancy must be estimated by patient's physician at > 6 months
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-3 (restricted to ECOG performance status [PS] 0-2 if age > 70 years)
* Patient must NOT have a history of allergic reaction attributable to compounds of similar chemical or biologic composition to 18F-FES
* Patient must NOT be in liver failure as judged by the patient's physician
* Histologically confirmed metastatic breast cancer
* Primary tumor and/or metastatic site must be ER+ and may be progesterone-receptor positive (PgR+) or progesterone-receptor negative (PgR-) by IHC; patients with a history of an estrogen-receptor negative (ER-) primary tumor and a documented ER+ metastatic site are eligible
* The pathology report and either (1) tissue (blocks or an unstained slides) or (2) a photomicrograph of the ER IHC slides from at least one site of metastatic disease and/or from primary breast cancer must be available for central review and analysis

  * NOTE: if photomicrographs are submitted, the submission of hematoxylin and eosin (H&E), PR and Ki67 IHC's, if performed, are also to be submitted
* Patient must NOT have human epidermal growth factor-2 positive (HER2+) metastatic disease
* Patient must NOT be planning to receive molecular targeted therapy (such as everolimus or palbociclib) nor HER2 directed therapy in addition to endocrine therapy
* Patient must NOT have received prior endocrine therapy for metastatic disease (i.e., must be first-line endocrine therapy for metastatic disease)
* Patient is not now, and never has received adjuvant endocrine therapy OR patient is currently receiving or has received adjuvant endocrine therapy in the past, AND adjuvant endocrine therapy was initiated > 2 years prior to diagnosis of metastatic disease

  * Note: patients who developed metastatic disease while still receiving adjuvant endocrine therapy must have a planned change in the type of endocrine agent used for subsequent metastatic disease treatment; patient is not receiving blocking adjuvant therapy (such as toremifene or tamoxifen) OR patient is receiving blocking adjuvant therapy, but will stop this therapy a minimum of 60 days prior to FES-PET/CT while still complying with the study timeline
* Patient must NOT have a history of > 1 line of administered chemotherapy for metastatic disease and must be off chemotherapy for a minimum of 2 weeks; prior chemotherapy in the adjuvant setting is allowed
* Disease may be measurable (by Response Evaluation Criteria in Solid Tumors [RECIST] 1.1 criteria) or non-measurable but must be present in at least one non-liver site, where presence is defined as 1.5 cm or greater and visualized on PET/CT with [18F]-fluorodeoxyglucose (FDG); patients with effusion only disease or disease only in the liver are not eligible for the study
* Patient must be able to lie still for a 20-30 minute PET/CT scan
* Patient must NOT weigh more than the maximum weight limit for the table for the PET/CT scanner at the institution where the study is being performed
* The patient is participating in the trial at an institution which has agreed to perform the imaging research studies, completed the ECOG-American College of Radiology Imaging Network (ACRIN) defined scanner qualification procedures and received ECOG-ACRIN (or current ACRIN) approval

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2016-05-04 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Negative predictive value of 18F FES uptake for response (CB), defined as the proportion of patients with a negative FES test result who have progressive disease | At 6 months
  FES-PET results will be assessed as positive or negative by quantitative or qualitative criteria. FES SUVmax < 1.5 will be defined as quantitatively negative test result while one or more sites of active disease will be qualitatively negative test result. The reference standard is patient's tumor response categorized by either CB or PD at 6 months. As part of the preliminary analysis, rates of FES uptake negative results overall and next by tumor response status will be calculated. FES-PET test positive results will be compared in the two tumor response groups using a chi-square test.

SECONDARY OUTCOMES:
Test-retest reproducibility of quantitative assessment of tumor FES uptake by SUVs | Up to 6 months
  The reproducibility of the two measurements of SUVs will be assessed by intra-class correlation coefficient and its 95% confidence interval (CI). Additionally, the coefficient of repeatability (CR) and the Bland-Altman plot will be used.
FES SUVmax | Up to 6 months
  The receiver operating characteristic (ROC) curve of FES SUVmax and its associated area under an ROC curve (AUC) will be estimated to predict tumor response (clinical benefit). Next, sensitivity and specificity of the dichotomized FES SUVmax (using a cutoff of 1.5) will be estimated non-parametrically, where sensitivity is the proportion of responders having FES SUVmax < 1.5 and specificity is the proportion of non-responders having FES SUVmax > 1.5.
Predictive accuracy of FES PET/CT for PFS, defined as the time from entry onto study until tumor progression or death from any cause | Up to 1 year
  To evaluate the predictive accuracy of FES PET, the time-dependent ROC curve of FES SUVmax at pre-specified time points (e.g. 6 months, 1 year) and its corresponding AUC will be estimated. Next, sensitivity and specificity of the dichotomized FES SUVmax (using a cutoff of 1.5) will be estimated in which reference standard is PFS status at pre-specified time points including 6 months and 1 year.
Significance of FES PET measures in predicting PD or CB, in concert with semi-quantitative interpretation of ER, PgR, and Ki-67 | Baseline
  Logistic regression analysis will be used to examine the effects of various FES PET measurements on clinical benefit. Predictors are semi-quantitative ER measure, PgR, and Ki-67 based on IHC. Significance of each FES PET measure will be determined by the odds ratio and its 95% CI.
FES uptake, as measured by SUVmax and semi-quantitative ER from IHC | Up to 6 months
  The semi-quantitative ER measure will be obtained by using Allred score. The relationship between SUVmax and semi-quantitative ER measure will be evaluated by using a linear regression model treating SUVmax as a dependent variable and semi-quantitative ER measure as a predictor.
FES SUVmax < 1.5 as the optimal cutpoint for predicting PFS | Up to 1 year
  Time dependent ROC analysis will be performed to determine the optimal cutoff point for the FES SUVmax and to examine whether there is a more optimal cut-off for dichotomous interpretation of FES SUVmax than the current value 1.5. Specifically, the optimal cut-off point will be determined by maximizing Youden's index for the time dependent ROC curve at a pre-specified time point (e.g. 6 months, 1 year).
Percent of eligible patients for whom biopsy is not feasible, i.e., clinical utility of indirect assay of ER expression by FES PET | Up to 6 months
  The proportion of eligible patients for whom biopsy of a metastatic site is not feasible out of a total of 99 patients will be calculated.
Heterogeneity of tumor FES uptake in individual patients defined as variability in lesion's FES uptake | Up to 6 months
  Sample correlation matrix for the multiple SUV measurements will be calculated. Next, linear mixed effects model will be used where the outcome is SUV measurements and covariates include fixed effects (sites that the SUV value is measured and patient characteristics). Lesion-specific random effects will be added to the model. The correlations among SUV measurements will be calculated based on the fitted model.

CONTACTS AND LOCATIONS:
Overall Officials: Farrokh Dehdashti, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (25):
- United States (25):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Springmill Medical Center, Indianapolis, Indiana
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Mount Sinai Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Fox Chase Cancer Center - East Norriton Hospital Outpatient Center, East Norriton, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin